CLINICAL TRIAL: NCT06060886
Title: Open-label, Multicenter, Randomized Clinical Trial to Evaluate the Efficacy and Safety of Aripiprazole vs Paliperidone/Risperidone Using Multi-omics Data in Patients With a First Episode Psychosis
Brief Title: Multidisciplinary Design to Optimize Schizophrenia Treatment Based on Multi-omics Data and Systems Biology Analysis
Acronym: SchizOMICS
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Consorcio Centro de Investigación Biomédica en Red (CIBER) (Other Government)
Collaborators: Instituto de Salud Carlos III (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SchizOMICS
Record Dates: First submitted 2023-05-16; First posted 2023-09-29 (Actual); Last update posted 2023-09-29 (Actual); Status verified 2023-06

CONDITIONS: Schizophrenia; Treatment-resistant Schizophrenia; Side Effect; Lipid Metabolism Disorders; Diabetes; NAFLD; Psychosis
MeSH Terms: conditions — Schizophrenia; Schizophrenia, Treatment-Resistant; Lipid Metabolism Disorders; Diabetes Mellitus; Non-alcoholic Fatty Liver Disease; Psychotic Disorders | interventions — Aripiprazole; Paliperidone Palmitate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- First episode of psychosis patients (Experimental): Operational definition for a "first episode of psychosis" included individuals with a non-affective psychosis who have not received previous antipsychotic treatment regardless of the duration of psychosis.
  Interventions: Drug: Aripiprazole; Drug: Paliperidone

INTERVENTIONS:
Drug: Aripiprazole — Oral dose range 5-30 mg/day (100 mg- 600 CPZeq). Long -acting injectables will be highly recommended in order to certify adherence.
Drug: Paliperidone — Oral dose range 3-12 mg/day (150mg-600 CPZeq). Long -acting injectables will be highly recommended in order to certify adherence

SUMMARY:
SchizOMICS is a Phase IV, multicenter, dose-flexible, open-label, randomized controlled clinical trial to evaluate the efficacy and safety of aripiprazole versus paliperidone using multi-omics data in patients with a first psychotic episode. The trial will include a total of 244 patients, with two arms of treatment with paliperidone and aripiprazole (1:1).

The main objectives of the study are:

1. To compare the efficacy and safety of aripiprazole and paliperidone in the treatment of first episode psychosis (FEP) subjects in real-world clinical settings at 3 months.
2. To elucidate whether non-responders after 3 months of adequate treatment may display different molecular signatures at baseline based on multi omics data and systems biology analysis.
3. To uncover whether the appearance of side effects after 1 year of adequate treatment may be related to different molecular signatures based on multi-omics data and lifestyle phenotype using systems biology analysis.

ELIGIBILITY:
Inclusion Criteria:

1. 15-40 years;
2. living in the catchment area;
3. experiencing a first episode of psychosis;
4. no prior treatment with antipsychotic medication or, if previously treated, a total lifetime of adequate antipsychotic treatment of less than 6 weeks;
5. Diagnostic and Statistical Manual of Mental Disorders fth Edition (DSM-5) criteria for schizophreniform disorder, schizophrenia, or schizoaffective disorder.

Exclusion Criteria:

1. meeting DSM-5 criteria for drug dependence;
2. meeting DSM-IV criteria for mental retardation;
3. having a history of neurological disease or head injury.

Ages: 15 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 244 (Estimated)
Dates: Start 2023-11-01 (Estimated); Primary Completion 2025-06-01 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Number of patients with a therapeutic response to aripiprazole or paliperidone | 3 months
  Considering response as a reduction in the Positive and Negative Symptom Scale (PANSS) > 50%.
  PANSS is a test made up of 30 items that are scored from 1 (absent) to 7 (extreme).
Number of patients with a therapeutic response to aripiprazole or paliperidone | 3 months
  Considering response as Clinical Global Impression severity scale for schizophrenia (ICG-ESQ-SI) < 4 points.
  ICG-ESQ-SI is a test made of 5 items that are scored from 1 (absent) to 7 (extreme).

SECONDARY OUTCOMES:
Number of patients with changes in negative symptoms | 12 months
  Using Scale for the Assessment of Negative Symptoms (SANS), test made of 25 items that are scored from 1 (absent) to 5 (extreme).
Number of patients with changes in depressive symptoms | 12 months
  Using Calgary Depression Scale for Schizophrenia (CDSS), test made of 9 items that are scored from 1 (absent) to 4 (extreme).
Number of patients with changes in functionality | 12 months
  Using Personal and Social Performance scale (PSP), test made of 4 items that are scored from 1 (absent) to 6 (extreme).
Number of patients with changes in quality of life | 12 months
  Using EuroQoL, test made of 1 item that are scored from 0 (worst) to 100 (best).
Number of patients with side effects | 12 months
  Using UKU Side Effect Rating Scale, test made of 56 items that are scored from 0 (absent) to 3 (extreme).

CONTACTS AND LOCATIONS:
Overall Officials: Javier Labad Arias, MD, PhD, Principal Investigator — Consorci Sanitari del Maresme, Hospital de Mataró

IPD SHARING:
Plan to Share IPD: No